CLINICAL TRIAL: NCT04779281
Title: Effects of Nutritional Status and Probiotics on Exercise-Related Clinical and Gastrointestinal Symptoms and Endurance Performance in Ultra-Endurance Athletes
Brief Title: Effects of Probiotics and Nutritional Status on Exercise-Induced Symptoms, and Endurance Performance in Ultra-Endurance Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Asli Devrim Lanpir, Research Assistant, PhD, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KA-180011; 18-AKD-89 (Other: Turkey Medicines and Medical Devices Agency)
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Ultra-endurance Athletes With Gastrointestinal Symptoms
Keywords: signs and symptoms, digestive; Probiotics; Oral rehydration therapy; Gastrointestinal Microbiome
MeSH Terms: conditions — Signs and Symptoms, Digestive

STUDY DESIGN:
Intervention Model Description: Ultra-endurance athletes with at least one gastrointestinal symptoms will be administered oral rehydration salts supplemented with L. Rhamnosus GG or oral rehydration salts only for 4 weeks
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Rehydration Salts supplemented with L. Rhamnosus GG (Experimental): a supplement containing sodium chloride, trisodium citrate, potassium chloride, dextrose, Lactobacillus Rhamnosus GG ATC53103 HN019 strain and fructooligosaccharides
  Interventions: Dietary Supplement: Oral Rehydration Salts only
- Oral Rehydration Salts only (Experimental): A supplement containing sodium chloride, trisodium citrate, potassium chloride, dextrose, microcrystalline cellulose
  Interventions: Dietary Supplement: Oral Rehydration Salts supplemented with L. Rhamnosus GG

INTERVENTIONS:
Dietary Supplement: Oral Rehydration Salts supplemented with L. Rhamnosus GG — A supplement containing sodium chloride, trisodium citrate, potassium chloride, dextrose, Lactobacillus Rhamnosus GG ATC53103 HN019 strain and fructooligosaccharides
  Arms: Oral Rehydration Salts only
Dietary Supplement: Oral Rehydration Salts only — A supplement containing sodium chloride, trisodium citrate, potassium chloride, dextrose, microcrystalline cellulose
  Arms: Oral Rehydration Salts supplemented with L. Rhamnosus GG

SUMMARY:
Ultra-endurance athletes have been commonly endured extreme conditions during races and training sessions, resulting in exercise-associated clinical symptoms, including gastrointestinal symptoms, dehydration, and elevated oxidative stress. Although these alterations adversely affect sports performance and well-being, there is no certain treatment or consensus on alleviating the exercise-associated clinical symptoms in ultra-endurance athletes. The objective of this study is to determine the effects of oral rehydration salts supplemented with Lactobacillus Rhamnosus GG on exercise-induced gastrointestinal problems, dehydration and oxidative stress in ultra-endurance athletes. Additionally, we aimed to assess the exercise-induced alterations in oxidative stress determined by applying an acute strenuous exercise protocol ((a cycle ergometer (45 min at 65%VO2max) immediately followed by a treadmill test (75% VO2max to exhaustion)) before and after the supplementation period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who train at least 15 h per week,
* Participants who do not have any metabolic disease,
* Have had at least one gastrointestinal symptom determined by using a Gastrointestinal Symptoms Rating Scale and Bristol Stool Chart Form Scale,
* Being a non-smoker,
* Have participated in at least one ultra-endurance race/event (lasts > 4 hr),
* Taking no vitamins, minerals, dietary supplements, antibiotics, and any medication at least during the three months before the study,
* (For women) participants with a regular menstrual cycle of physiological length (24-35 days)

Exclusion Criteria:

* Regular tobacco use
* Inability to adhere to any of the study protocol requirements (i.e. alcohol, caffeine consumption, diet control)
* Having consumed any supplements and/or medicines for the preceding 3 months period.
* (For women) participants in menopause or using oral contraceptives

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Changes of the gut microbiome after a 4-week supplementation period | Change from Baseline Gut Microbiome at 4 weeks
  - To assess the profile of gut flora (% abundance of various bacterial phyla, families, genera and species) at baseline and after supplementation in ultra-endurance athletes, using a 16S ribosomal RNA sequencing

SECONDARY OUTCOMES:
Changes in blood markers of exercise-associated oxidative stress (8-isoprostaglandin 2Fa, Total Antioxidant Capacity, and Total Oxidant Capacity in plasma) | 4 weeks
  - Blood samples were collected pre-and post-exercise applied before and after supplementation to evaluate the change in exercise-induced oxidative stress in plasma. Plasma concentrations of 8-isoprostaglandin 2Fa, Total Antioxidant Capacity, and Total Oxidant Capacity were analysed using ELISA kits.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğba Kocahan, MD, Study Director — Centre of Athlete Training and Health Research
Locations (1):
- Centre of Athlete Training and Health Research, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krabak BJ, Lipman GS, Waite BL, Rundell SD. Exercise-Associated Hyponatremia, Hypernatremia, and Hydration Status in Multistage Ultramarathons. Wilderness Environ Med. 2017 Dec;28(4):291-298. doi: 10.1016/j.wem.2017.05.008. Epub 2017 Aug 7. PMID 28781178
- [Result] Nocella C, Cammisotto V, Pigozzi F, Borrione P, Fossati C, D'Amico A, Cangemi R, Peruzzi M, Gobbi G, Ettorre E, Frati G, Cavarretta E, Carnevale R; SMiLe Group. Impairment between Oxidant and Antioxidant Systems: Short- and Long-term Implications for Athletes' Health. Nutrients. 2019 Jun 15;11(6):1353. doi: 10.3390/nu11061353. PMID 31208096
- [Result] Pyne DB. Exercise-induced muscle damage and inflammation: a review. Aust J Sci Med Sport. 1994 Sep-Dec;26(3-4):49-58. PMID 8665277
- [Result] Lopez AA, Preziosi JP, Chateau P, Auguste P, Plique O. [Digestive disorders and self medication observed during a competition in endurance athletes. Prospective epidemiological study during a championship of triathlon]. Gastroenterol Clin Biol. 1994;18(4):317-22. French. PMID 7958646
- [Result] Maughan RJ, Shirreffs SM. Sports Beverages for Optimizing Physical Performance. In: Wilson T., Temple N. (eds) Beverage Impacts on Health and Nutrition. Nutrition and Health. Humana Press, Cham. 2016.
- [Result] Mach N, Fuster-Botella D. Endurance exercise and gut microbiota: A review. J Sport Health Sci. 2017 Jun;6(2):179-197. doi: 10.1016/j.jshs.2016.05.001. Epub 2016 May 10. PMID 30356594
- [Result] Hoffman MD, Stellingwerff T, Costa RJS. Considerations for ultra-endurance activities: part 2 - hydration. Res Sports Med. 2019 Apr-Jun;27(2):182-194. doi: 10.1080/15438627.2018.1502189. Epub 2018 Jul 28. PMID 30056755
- [Result] Hooper LV, Gordon JI. Commensal host-bacterial relationships in the gut. Science. 2001 May 11;292(5519):1115-8. doi: 10.1126/science.1058709. PMID 11352068
- [Result] Kekkonen RA, Vasankari TJ, Vuorimaa T, Haahtela T, Julkunen I, Korpela R. The effect of probiotics on respiratory infections and gastrointestinal symptoms during training in marathon runners. Int J Sport Nutr Exerc Metab. 2007 Aug;17(4):352-63. doi: 10.1123/ijsnem.17.4.352. PMID 17962710
- [Result] Martarelli D, Verdenelli MC, Scuri S, Cocchioni M, Silvi S, Cecchini C, Pompei P. Effect of a probiotic intake on oxidant and antioxidant parameters in plasma of athletes during intense exercise training. Curr Microbiol. 2011 Jun;62(6):1689-96. doi: 10.1007/s00284-011-9915-3. Epub 2011 Mar 12. PMID 21400082